CLINICAL TRIAL: NCT06866535
Title: VIP - Vascular Infection Project : Prospective Multicentric Database on Vascular Infections
Brief Title: VIP - Vascular Infection Project
Acronym: Cohorte VIP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/01
Record Dates: First submitted 2024-06-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Aortitis; Vascular Graft Infection; Blood Vessel Prosthesis; Infections
Keywords: vascular graft and endograft infections; infectious aortitis; infectious arteritis
MeSH Terms: conditions — Aortitis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Native vascular infection
- Prosthetic vascular infections

SUMMARY:
Constitution of a prospective multicentric observational database to study vascular infections, both native, especially aortitis, and vascular graft and endograft infections. Clinical and paraclinical data on medical, surgical, anesthetic and intensive care management will be collected in order to better characterize these infections

DETAILED DESCRIPTION:
Vascular infections are rare but severe, burdened by high morbi-mortality and recurrence rates. However, many questions remain regarding their management which is still not consensual, both surgical and medical management. The term "vascular infections" encompasses vascular graft and endograft infections, as well as infections of native arteries and the aorta. For vascular graft infections, the optimal surgery is to remove the infected graft before vascular reconstruction with a new graft, either synthetic or biologic. However, some patients are too fragile to undergo surgery and might then benefit from an endovascular graft, an abscess drainage or no surgery at all, only medical treatment. For native arterial infections, surgery is often required to remove the infected arterial wall before vascular reconstruction. However, some patients cannot be operated on and might also benefit from an endovascular surgery. In these two vascular infections, the ideal anti-microbial treatment is uncertain, whether it pertains to the duration of therapy, the type of molecules, or their number. All of these medical and surgical factors may impact the prognosis of patients and should be collectively assessed in order to determine the best strategy for enhancing their outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years-old;
* all patients with a vascular infection, either native (aortitis, arteritis) or prosthetic (vascular graft, endograft and/or stent),
* oral consent

Exclusion Criteria:

* patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ents with a vascular infection, either native (aortitis, arteritis) or prosthetic (vascular graft, endograft and/or stent)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2032-05-10 (Estimated); Study Completion 2032-05-10 (Estimated)

PRIMARY OUTCOMES:
mortality | Year 1
  mortality r

SECONDARY OUTCOMES:
mortality | Day 30, Year 2, Year 5
  mortality rate
morbidity | Year 1
  morbidity rate
relapse | year 1, Year 2, Year 5
  relapse rates
reinfection | year 1, Year 2, Year 5
  reinfection rates

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France